CLINICAL TRIAL: NCT00258466
Title: Phase III Trial of Neutron + Photon Radiation Versus Photon + Hypofractionated Intensity Modulated Radiation Therapy in Localized Prostate Cancer
Brief Title: Radiation Therapy in Treating Patients With Stage I, Stage II, or Stage III Prostate Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000447161; P30CA022453 (NIH); WSU-D-2879; WSU-HIC-047405MP4F
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Giving radiation therapy in different ways may kill more tumor cells. It is not yet known which type of radiation therapy is more effective in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying different types of radiation therapy to compare how well they work in treating patients with stage I, stage II, or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of neutron and photon radiotherapy vs hypofractionated intensity modulated radiation, in terms of a lower frequency of chronic complication rate (chronic toxicity and disease-free survival), in patients with favorable to intermediate prognosis, stage I-III adenocarcinoma of the prostate.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to stage of disease (T1 vs T2 vs T3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo neutron radiotherapy over 15-45 minutes 5 days a week for 2 weeks followed by photon radiotherapy over 15-45 minutes 5 days a week for 5 weeks.
* Arm II: Patients undergo photon radiotherapy over 15-45 minutes 5 days a week for 5 weeks followed by hypofractionated photon irradiation over 15-45 minutes 5 days a week for 2 weeks.

After completion of study treatment, patients are followed periodically for 5 years and then yearly thereafter.

PROJECTED ACCRUAL: A total of 300 patients (150 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Stage I-III disease (T1-T3, N0, M0)
  * No clinical or radiographic evidence of metastasis

    * If prostate-specific antigen (PSA) ≥ 10.0 ng/mL and Gleason score is 7, a radioisotope bone scan must show no evidence of metastasis
    * No evidence of lymphatic or visceral metastases of the abdomen or pelvis on CT scan or MRI
* PSA ≤ 20 ng/mL
* Gleason score ≤ 7 (if stage T3 , score must be < 7)

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* More than 10 years

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Endocrine therapy

* Prior hormonal therapy allowed provided it was initiated no more than 2 months ago, and may include the following:

  * Luteinizing hormone-releasing hormone agonists (e.g., goserelin, leuprolide)
  * Anti-androgens (e.g., flutamide, bicalutamide)

Radiotherapy

* No prior pelvic irradiation

Surgery

* No prior radical prostatectomy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of chronic grade 2 or higher toxicity as measured by RTOG/EORTC late morbidity scoring scheme at 1, 4, 8, and 12 months after treatment, then every 6 months for 5 years, then annually

SECONDARY OUTCOMES:
Disease free survival at 1, 4, 8, and 12 months after treatment, then every 6 months for 5 years, then annually

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D. Forman, MD, FACR, Study Chair — Weisberg Cancer Treatment Center